CLINICAL TRIAL: NCT07194694
Title: Dexmedetomidine vs Ketamine as Adjuvants to Bupivacaine in Transversus Abdominus Plane Block in Inguinal Hernioplasty: A Randomized Clincal Controlled Trial
Brief Title: Dexmedetomidine vs Ketamine as Adjuvants to Bupivacaine in Transversus Abdominus Plane Block in Inguinal Hernioplasty
Acronym: DEX\KET in TAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Mikhail Fouad Hanna, Assistant Lecturer at Department: Anesthesiology, Intensive Care and Pain Management, Faculty of Medicine, Ain Shams University., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD 42
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Relief
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Ketamine

STUDY DESIGN:
Intervention Model Description: At the end of surgery an ipsilateral US guided TAP block (posterior approach) will be given to all the patients by placing linear US probe (high frequency probe 10-12 MHz) connected to a portable US unit initially in the mid-axillary plane midway between the lower costal margin and the highest point of iliac crest, then it will be moved posteriorly till a scan reveals the transversus abdominis muscle tailing off into the aponeurosis, near the Quadratus lumborum muscle. The injection site is superficial to the aponeurosis near quadratus lumborum. while the patient in supine position with slight lateralization After skin disinfection, a 22-G needle with an injection line will be inserted in plane with the probe. Once the tip of the needle is placed in place and after negative suction 5 ml saline 0.9% will be injected to verify the right place, then one of the three study solutions will be injected.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sampling Method: Simple random sample. Randomization: Computer generated random list. Blinding: The patient, the physician performing the block and the investigator will be blinded as regard tools and patient's group.
  Concealment: Randomization list will be concealed from all members off the study, known only by one person which is not included in it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DEX on TAP (Active Comparator): Group A (Dexmedetomidine Group): patients will receive 20 ml solution containing 1 mg/kg bupivacaine + 1mcg/kg dexmedetomidine +normal saline.
  Interventions: Drug: Dexmedetomidine & Bupivacaine.
- KET on TAP (Active Comparator): Group B (ketamine Group): patients will receive 20 ml solution containing 1 mg/kg bupivacaine+0.5 mg/kg ketamine + normal saline.
  Interventions: Drug: ketamine and bupivacaine injection
- TAP (Placebo Comparator): Group C (Control Group): Patients will receive 20 ml solution containing 1 mg/kg bupivacaine + normal saline.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine & Bupivacaine. — Group A (Dexmedetomidine Group): patients will receive 20 ml solution containing 1 mg/kg bupivacaine + 1mcg/kg dexmedetomidine +normal saline.
  Arms: DEX on TAP
Drug: ketamine and bupivacaine injection — Group B (ketamine Group): patients will receive 20 ml solution containing 1 mg/kg bupivacaine+0.5 mg/kg ketamine + normal saline.
  Arms: KET on TAP
Drug: Bupivacaine — Group C (Control Group): Patients will receive 20 ml solution containing 1 mg/kg bupivacaine + normal saline.
  Arms: TAP

SUMMARY:
This clinical trial aims to compare the effect of adding dexmedetomidine versus ketamine to bupivacaine in transversus abdominis plane block in patients undergoing unilateral inguinal hernioplasty. The key questions it is expected to answer are:

To what extent do dexmedetomidine and ketamine adjuvants, when combined with bupivacaine, offer a longer analgesic period in a Transversus Abdominis Plane (TAP) block?

To investigate the pain at rest and coughing with particular time intervals (0, 2, 4, 6, and 12 hours) after the operation.

researchers will rely on three groups:

Group A (Dexmedetomidine Group): patients will receive 20 ml solution containing 1 mg/kg bupivacaine + 1 mcg/kg dexmedetomidine + normal saline.

Group B (ketamine group): patients will receive 20 ml of solution containing 1 mg/kg bupivacaine + 0.5 mg/kg ketamine + normal saline.

Group C (Control Group): Patients will receive 20 ml of solution containing 1 mg/kg bupivacaine + normal saline.

Participants will:

have general anesthesia in their planned unilateral hernioplasty. have an ipsilateral US guided TAP block (posterior approach) using one of the three study solutions at the end of the surgery prior to be waked up.

Measure their Numeric Pain Rating Scale (NRS) at rest and coughing at particular time intervals (0, 2, 4, 6, and 12 hours) after the operation.

DETAILED DESCRIPTION:
Preoperative Assessment:

Patients scheduled for unilateral inguinal hernioplasty will be assessed preoperatively by evaluating their medical history, laboratory investigations, and fulfillment of the above inclusion criteria. The patient's preparation will be done by IV cannulation with an 18G cannula, and infusion of 500 ml of Ringer's solution will be started, and about 20 minutes before anesthesia induction, midazolam (0.05 mg/kg) will be received as a sedative premedication.

Intraoperative Procedures and Assessments:

After reaching the operating room, standard monitoring will be applied, which includes electrocardiography (ECG), non-invasive blood pressure, and pulse oximetry for peripheral oxygen saturation (SPO2). After preoxygenation, induction of general anesthesia will be done by IV injection of propofol (2 mg/kg), fentanyl (2 mcg/kg), atracurium (0.5 mg/kg), and inhalational isoflurane 1.2%, followed by endotracheal intubation and controlled mechanical ventilation with tidal volume 7-8 ml/kg, respiratory rate 12/min, and FIO₂ 100%. Then anesthesia will be maintained by inhalational isoflurane, atracurium 0.1 mg/kg every 20 minutes, and intraoperative fluid (Ringer's solution), which was calculated to cover the maintenance, deficit, and 3rd space requirement.

At the end of surgery an ipsilateral US-guided TAP block will be given to all the patients by placing a linear US probe (high-frequency probe 10-12 MHz) connected to a portable US unit initially in the mid-axillary plane midway between the lower costal margin and the highest point of iliac crest, then it was moved posteriorly till a scan reveals the transversus abdominis muscle tailing off into the aponeurosis, near the Quadratus lumborum muscle. The injection site was superficial to the aponeurosis near quadratus lumborum. while the patient in supine position with slight lateralization After skin disinfection, a 22-G needle with an injection line will be inserted in plane with the probe. Once the tip of the needle is placed in place, and after negative suction, 5 ml of 0.9% saline will be injected to verify the right place, then one of the three study solutions will be injected.

Group A (Dexmedetomidine Group): patients received 20 ml solution containing 1 mg/kg bupivacaine + 1 mcg/kg dexmedetomidine + normal saline.

Group B (Ketamine Group): patients received 20 ml solution containing 1 mg/kg bupivacaine + 0.5 mg/kg ketamine + normal saline.

Group C (Control Group): Patients received 20 ml of solution containing 1 mg/kg bupivacaine + normal saline.

Then discontinuation of inhalational isoflurane and reversal of muscle blockade by a neostigmine 0.05 mg/kg and atropine (0.01-0.02 mg/kg) mixture, and after fulfillment of extubation criteria, extubation was done.

Postoperative analgesic regimen:

When NRS >3: Nalbuphine (0.1 mg/kg) will be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral inguinal hernioplasty of ASA I or II.
* Age group: 18-60 years old.

Exclusion Criteria:

* Patient refusal.
* known allergy to any of the used drugs
* ASA III or above
* Coagulation disorders and thrombocytopenia
* Body mass index (BMI) >30
* Infection at needle insertion site
* Patients undergoing bilateral inguinal hernioplasty

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale | Immediately postoperative - 2 hours postoperatively - 4 hours postoperatively - 6 hours postoperatively - 12 hours postoperatively
  The Numeric Pain Rating Scale (NRS) is an effective method for measuring pain intensity. It consists of an 11-point scale where:
  0 represents no pain - 10 represents the worst pain imaginable. Patients are asked to select a whole number that best reflects their pain intensity or average pain level.

SECONDARY OUTCOMES:
Change in Mean arterial blood pressure | Immediately postoperative - 2 hours postoperative - 4 hours postoperative
  MAP = Diastolic Blood Pressure + (1/3 * Pulse Pressure). It is the average pressure in your arteries throughout one cardiac cycle and will be calculated after measuring the blood pressure of the patients postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No